CLINICAL TRIAL: NCT04420429
Title: The Effect Of Preoperative Anterior Segment Parameters On Success After Descemet Membrane Endothelial Keratoplasty (Dmek) Surgery
Brief Title: The Effect Of Preoperative Parameters On Success After DMEK Surgery
Status: Completed | Type: Observational
Sponsor: Beyoglu Eye Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Semih Çakmak, Principal Investigator, Beyoglu Eye Research and Education Hospital
Other Study IDs: BeyogluEREH
Record Dates: First submitted 2020-05-16; First posted 2020-06-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Fuchs' Endothelial Dystrophy; Pseudophakic Bullous Keratopathy; Descemet's Membrane; Defect; Herpetic Keratitis; Angle's Classification; Endothelial Dysfunction
Keywords: Descemet Membrane; anterior chamber depth; axial length; endothelial count; Descemet membrane endothelial keratoplasty
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Keratitis, Herpetic; Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: All patients
  Interventions: Procedure: Descemet membrane endothelial keratoplasty (DMEK)

INTERVENTIONS:
Procedure: Descemet membrane endothelial keratoplasty (DMEK) — All participants underwent DMEK surgery

SUMMARY:
The aim of this study is to evaluate the effect of preoperative parameters on surgical results in Descemet Membrane Endothelial Keratoplasty (DMEK) surgery.

DETAILED DESCRIPTION:
In patients undergoing Descemet Membrane Endothelial Keratoplasty (DMEK) surgery; preoperative anterior chamber depth, angle parameters, axial length and corneal parameters will be evaluated. The effects of these parameters on surgical results will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo Descemet membrane endothelial keratoplasty(DMEK)
* aged 18 old older

Exclusion Criteria:

* Patients with corneal pathology other than endothelial insufficiency
* Glaucoma patients,
* Patients who have previously had any keratoplasty procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who developed pseudophakic bullous keratopathy, Fuchs endothelial dystrophy, endothelial insufficiency after herpetic endotheliitis and associated permanent corneal edema and therefore DMEK surgery.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity | Baseline and after surgery 1, 3, 6, and 12 months
  Change from baseline
Change in endothelial cell density | after surgery 1, 3, 6, and 12 months
  Change from baseline

SECONDARY OUTCOMES:
Change in maximum (steepest) and minimum (flattest) keratometry values in the central corneal zone | Baseline and after surgery 1, 3, 6, and 12 months
  Change from baseline
Change in anterior chamber depth | Baseline and after surgery 1, 3, 6, and 12 months
  Change from baseline
Change in axial length | Baseline and after surgery 1, 3, 6, and 12 months
  Change from baseline
Change in central pachymetry | Baseline and after surgery 1, 3, 6, and 12 months
  Change from baseline
Change in intraocular pressure | Baseline and after surgery 1, 3, 6, and 12 months
  Change from baseline

OTHER OUTCOMES:
Surgical complications | During surgery
  Complications occurring during the surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Çakmak, MD, Principal Investigator — Beyoglu Eye Training and Research Hospital
Locations (1):
- Beyoğlu Eye Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cakmak S, Kirgiz A, Yildirim Y, Taskoparan S, Genc S, Agca A. The effect of anterior segment parameters on surgical success of Descemet membrane endothelial keratoplasty: a prospective study. Int Ophthalmol. 2023 Jan;43(1):197-205. doi: 10.1007/s10792-022-02416-0. Epub 2022 Jul 10. PMID 35810243

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT04420429/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT04420429/ICF_001.pdf